CLINICAL TRIAL: NCT00685971
Title: Randomized Placebo-Controlled Trial of Cholecalciferol for Vitamin D Deficiency in Adults With Cystic Fibrosis
Brief Title: Cholecalciferol for Vitamin D in Adult Cystic Fibrosis (CF) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMH 07-036
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2011-07

CONDITIONS: Cystic Fibrosis; Vitamin D Deficiency
Keywords: Cystic Fibrosis; Vitamin D deficiency
MeSH Terms: conditions — Cystic Fibrosis; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): vitamin
  Interventions: Dietary Supplement: 5000 IU of cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: 5000 IU of cholecalciferol — 5 drops taken once daily for 12 weeks
  Arms: Vitamin D
Dietary Supplement: placebo — 5 drops once daily for 12 weeks
  Arms: Placebo

SUMMARY:
The main aim of the research question to test the primary hypothesis of this study, namely, Does 12 weeks of an additional 5000 IU daily of cholecalciferol increase serum 25OHD levels in adults with Cystic Fibrosis (CF) who have vitamin D deficiency relative to placebo?

DETAILED DESCRIPTION:
Background and Significance Vitamin D is a fat-soluble vitamin necessary to maintain bone health as it maximizes calcium absorption from the gastrointestinal tract. Our primary source of vitamin D is through skin synthesis following exposure to solar UV-B irradiation. Natural dietary sources are limited which has led to the fortification of milk and baby formula with vitamin D.1 Vitamin D deficiency reduces dietary calcium absorption to 10-15% whereas 30 to 40% is absorbed when vitamin D levels are adequate.2 Although the effect of vitamin D is primarily on calcium homeostasis, vitamin D receptors can be found on many different cells within the body suggesting vitamin D has an impact beyond bones. Several epidemiological studies have shown an association between vitamin D and the prevalence of multiple sclerosis3, type 1 diabetes4;5, and cancer6. More recently, low vitamin D has been associated with lower lung function7;8 raising the possibility that vitamin D may influence pulmonary status. The active metabolite, 1,25 dihydroxyvitamin D, has a number of actions that may be relevant to respiratory diseases. It inhibits the formation of matrix metalloproteinases, inhibits fibroblast proliferations and influences collagen synthesis, all of which could influence tissue remodelling in the pulmonary airways.

Vitamin D deficiency: Definitions Vitamin D adequacy is traditionally assessed using circulating serum 25-hydroxyvitamin D (25OHD) levels. Concentrations below 25 nmol/L are associated with rickets and histologically evident osteomalacia indicating severe deficiency. Levels between 25 and 50 nmol/L are indicative of moderate deficiency and have been associated with mild elevations in parathyroid hormone(PTH) levels.9 However, there is a growing body of literature to suggest that levels below 75 nmol/L are inadequate. For example, healthy individuals on no vitamin D supplementation who live and work in sun-rich environments (i.e. lifeguards) have 25OHD levels between 100 and 158 nmol/L.10 Furthermore, vitamin D supplementation reduces fracture rates and improves bone mineral density (BMD) when serum 25OHD levels are > 100 nmol/L.11;12 And finally, 25OHD levels between 75 and 100 nmol/L result in maximal suppression of PTH and maximize calcium absorption from the gastrointestinal tract.13;14 This evidence supports the notion that the ideal target serum 25OHD level approximates 75 nmol/L or higher.

Vitamin D deficiency in Cystic Fibrosis Despite routine supplementation, the prevalence of vitamin D deficiency in cystic fibrosis (CF) is common ranging from 20 to over 80%, depending on the definition used to categorize the normal range.15-20 The etiology of low vitamin D in CF is poorly understood but contributing factors include decreased gastrointestinal absorption, impaired hydroxylation of vitamin D21, reduced sun exposure combined with increased use of sunscreens, seasonal influence as well as geographical location. Low bone mineral density has been well documented in CF and although bone disease in CF is likely multifactorial, vitamin D deficiency has been implicated as an etiologic factor15;17;19;22. Although few studies show a clear relationship between vitamin D and low bone density, it is plausible that sub-optimal serum vitamin D levels may aggravate bone disease in this population and that normalizing levels will maximize bone health. Furthermore, fracture risk appears to be increased in the CF population17;19;23. Vitamin D supplementation in elderly and osteoporotic subjects has been shown to reduce fractures, improve BMD and decrease falls11 but there are few studies examining the effect of vitamin D supplementation in CF16;18;24.

Treatment of vitamin D deficiency in CF Several forms of vitamin D supplementation have been used in an attempt to improve calcium homeostasis and normalize serum vitamin D levels in CF including cholecalciferol (animal form), ergocalciferol (plant form), and calcitriol (active 1,25-dihydroxyvitamin D). Which form of vitamin D and how much is needed to normalize serum levels most effectively in CF is unknown. Hanly et al assessed the response to 800 IU daily of cholecalciferol for a minimum of 4 weeks in twenty adolescents and young adults with CF. Serum levels of 25OHD increased although several subjects remained below the normal range despite supplementation.16 In the only published randomized placebo-controlled trial, Haworth et al studied 30 adults with CF and showed that calcium and cholecalciferol supplementation reduced the rate of bone turnover and bone loss although this did not reach statistical significance. Interestingly however, serum 25OHD levels were unchanged despite an additional 800 IU of cholecalciferol daily for 12 months.24 Pilot work recently published on our CF population shows that additional cholecalciferol can successfully increased serum 25OHD levels.25 This study was a retrospective review and a randomized clinical trial is needed to confirm these results. With ergocalciferol, Lark et al found absorption to be significantly lower and highly variable in adults with CF compared to controls.26 Furthermore, these patients demonstrated poor conversion of ergocalciferol to 25OHD raising the possibility of impaired hydroxylation by the hepatic enzyme, 25-hydroxylase. In 2005, Boyle et al showed that even with high-dose ergocalciferol (50-100,000 IU weekly), serum levels did not correct vitamin D deficiency to the target level of 75 nmol/L in subjects with CF.18 Some studies have shown that cholecalciferol is more efficacious than ergocalciferol in correcting vitamin D deficiency in the non-CF population.27;28 Possible mechanisms for this differential response to supplemental vitamin D include differences in affinity of vitamin D-binding protein for the two calciferols or increased affinity for the hepatic 25-hydroxylase for cholecalciferol. Finally, one study published showed short-term use of calcitriol, (1,25 dihydroxyvitamin D) increased calcium absorption in CF but serum 25OHD levels remained unchanged.29

In summary, there are many studies documenting vitamin D deficiency in the CF population however there is a paucity of literature evaluating treatment regimens to correct this deficiency. One may ask why not study a more clinically relevant outcome such as fracture rate or change in bone mineral density rather than a biochemical marker. Although these are definitely important clinical outcomes to examine, we feel that the CF population has unique factors that affect absorption of fats therefore it is difficult to estimate the amount of supplementation needed to achieve optimal serum levels (i.e. > 75 nmol/L) of 25OHD. Changes in serum levels can be seen within 4-8 weeks whereas changes in bone mineral density can take years to be detected. If vitamin D supplementation is inadequate to achieve optimal serum levels, changes in BMD and fractures may not be seen and the study results may be falsely negative. By determining the dosage required to achieve optimal serum levels first, this study will provide important information to researchers that can be used in long-term controlled clinical trials.

Research Question Aim The main aim of the research question to test the primary hypothesis of this study, namely, Does 12 weeks of an additional 5000 IU daily of cholecalciferol increase serum 25OHD levels in adults with CF who have vitamin D deficiency relative to placebo?

ELIGIBILITY:
Inclusion Criteria:

1. older than 18 years of age
2. diagnosis of CF by sweat testing/genetics
3. vitamin D deficiency defined as a serum 25OHD level < 75 nmol/L
4. on stable baseline vitamin D supplementation for at least 2 months. Standard vitamin D supplementation (cholecalciferol) in CF includes 800 IU daily for individuals with pancreatic insufficiency and 400 IU daily for those with pancreatic sufficiency

Exclusion Criteria:

1. Individuals with known hypercalcemia or renal stones
2. psychiatric history
3. use of tanning beds/travel to sunny location within the last 2 months
4. lung transplantation
5. pregnancy or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for this study is the change in mean serum 25OHD levels between the two groups | 12 weeks

SECONDARY OUTCOMES:
Mean change from baseline for pulmonary function testing (FEV1 and FVC) | 12 weeks
Mean change from baseline in serum calcium levels | 12 weeks
Mean change from baseline in parathyroid hormone levels | 12 weeks
Mean change from baseline in creatinine levels | 12 weeks
Change in the proportion of subjects whose 25OHD vitamin levels are above 75 nmol/L | 12 weeks
A subgroup analysis by pancreatic status will be done to assess the impact of this factor on serum 25OHD levels | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne Stephenson, Dr., Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada